CLINICAL TRIAL: NCT05233865
Title: Hemodynamic Effects During Land vs Water Exercise for Older Adults With Orthostatic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001869
Record Dates: First submitted 2021-10-21; First posted 2022-02-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water condition (Experimental): Participants blood pressure, heart rate and self-reported symptoms (such as dizziness) will be collected multiple times during sitting, standing and walking conditions when in a pool.
  Interventions: Behavioral: Water exercise
- Land condition (Active Comparator): Participants blood pressure, heart rate and self-reported symptoms (such as dizziness) will be collected multiple times during sitting, standing, and walking conditions when on land.
  Interventions: Behavioral: Land exercise

INTERVENTIONS:
Behavioral: Water exercise — Participants will be asked to sit and stand multiple times (before, immediately after, and 2 hours after a 15-minute walking session). The walking session will consist of 3 minutes of walking at a light intensity followed by 9 min of walking at a moderate intensity and a 3-minute cool down walking at a light intensity. This walking session will occur in a pool.
  Arms: Water condition
Behavioral: Land exercise — Participants will be asked to sit and stand multiple times (before, immediately after, and 2 hours after a 15-minute walking session). The walking session will consist of 3 minutes of walking at a light intensity followed by 9 min of walking at a moderate intensity and a 3-minute cool down walking at a light intensity. This walking session will occur on land.
  Arms: Land condition

SUMMARY:
The purpose of the study is to understand how blood pressure, heart rate, and symptoms of low blood pressure (such as dizziness or nausea) are affected by positional changes and exercise when on land or in the water for people who tend to experience orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of dizziness upon standing (from sit or supine position) or known diagnosis of orthostatic hypotension
* Able to stand independently for 3-5 consecutive minutes
* Able to walk independently (with or without an assistive devise)
* Medically stable for last month
* Score of 3 or greater on Mini-Cog (standardized outcome measure to detect dementia)
* Full coronavirus vaccination

Exclusion Criteria:

* Diagnosis of dementia
* Contraindication for pool exercise (such as infected open wounds, fecal incontinence, diarrhea.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) | <1 minute upon standing
  Blood pressure will be taken with an automated blood pressure device
Diastolic blood pressure (mmHg) | <1 minute upon standing
  Blood pressure will be taken with an automated blood pressure device
Self-reported orthostatic hypotension symptoms | 2 minutes
  A self-reported instrument assessing symptoms from low blood pressure experienced upon standing or after prolonged upright activities. Possible scores range from 0 (no symptoms) to 10 (worse possible symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Laboratory at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data available